CLINICAL TRIAL: NCT04851509
Title: Static Helical Screw Locking of Pertrochanteric Femur Fractures Using the TFN-Advanced Proximal Femoral Nailing System - a Randomized Trial
Brief Title: Static Helical Screw Locking of Pertrochanteric Femur Fractures Using the TFN-A
Acronym: TFN-A
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fraser Orthopaedic Research Society (Network)
Collaborators: DePuy Synthes (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FHREB#: 2021-015
Record Dates: First submitted 2021-04-14; First posted 2021-04-20 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Pertrochanteric Fracture

STUDY DESIGN:
Intervention Model Description: Randomized trial design utilizing alternating treatment allocation to assign patients to treatment arms, treatment allocations will last for two months at a time.
Who Masked: Participant, Outcomes Assessor
Masking Description: Surgeons cannot be blinded to the treatment allocation of the surgical intervention due to having to perform the static or dynamic rotational lock. Participants will be blinded to the form of locking they receive. Research personnel completing the outcome measures will be blinded. Data analyst(s) and the radiographic reviewer(s) will be blinded to the treatment arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dynamic rotational locking (Active Comparator): Using a fracture table, the affected leg will be placed into traction and the patient will be prepped and draped in the usual fashion. The fracture will be provisionally reduced using closed techniques. A 3cm incision will be used to gain access to the intramedullary canal and the nail (either a short nail or long nail, at the discretion of the treating surgeon) will be introduced to the femur. The screw will be placed across the fracture and into the femoral head, aiming for a tip-to-apex distance less than 25mm. The compression nut will be used to compress the fracture. The screw will be rotationally locked by using the 5mm hex flexible screwdriver by advancing the set screw until it stops completely. The screw will then be turned counterclockwise by a ½ turn.
  Interventions: Procedure: Dynamic Rotational Locking
- Static locking (Experimental): Using a fracture table, the affected leg will be placed into traction and the patient will be prepped and draped in the usual fashion. The fracture will be provisionally reduced using closed techniques. A 3cm incision will be used to gain access to the intramedullary canal and the nail (either a short nail or long nail, at the discretion of the treating surgeon) will be introduced to the femur. The screw will be placed across the fracture and into the femoral head, aiming for a tip-to-apex distance of less than 25mm. The compression nut will be used to compress the fracture. The screw will then be statically locked using the 6Nm torque-limiting blue handle with 6mm hex coupling to completely lock the set screw down on the helical screw.
  Interventions: Procedure: Static Locking

INTERVENTIONS:
Procedure: Dynamic Rotational Locking — Performed, as per the Synthes technique guide, using the 5mm hex flexible set screwdriver and then loosening the set screw by one-half turn of the screwdriver.
  Arms: Dynamic rotational locking
Procedure: Static Locking — Performed by using the torque-limiting set screwdriver and locking the set screw down onto the helical screw to prevent dynamic sliding of the screw within the nail.
  Arms: Static locking

SUMMARY:
The study will investigate the shortening and collapse of pertrochanteric fractures following surgical management with the TFN-Advanced nailing system. The focus will be on comparing radiographic assessments of nails which have been statically locked versus dynamically locked. This is a randomized control study with the initial invention being randomized to either statically locking or dynamically locking. For a two-month period, all eligible patients will receive the randomized allocated treatment, then treatment will switch to the alternate treatment for the next two months and will continue to alternate treatments for two-month periods until study enrollment has completed.

DETAILED DESCRIPTION:
Hip fractures are common injuries in the elderly population that result in significant morbidity and mortality and a significant burden on health care systems. Hip fractures can be treated with arthroplasty or with internal fixation, depending on the fracture pattern. Cephalomedullary nailing (CMN) has become one of the established treatments for intertrochanteric hip fractures with a wide variety of implant designs from many different companies. The TFN-ADVANCED™ Proximal femoral nailing system (TFN-A) is a novel implant for treating intertrochanteric and subtrochanteric proximal femur fractures with a paucity of published literature on the performance of this implant.

A method to decrease the amount of fracture compression is to use the set screw to lock the screw "statically" so it does not slide to the same degree as if the screw is placed in the "dynamic" or sliding position. To the knowledge of the investigators, the role of statically locking the screw to prevent fracture collapse has not been studied. Statically locking CMN to treat hip fractures has become standard of care at the Royal Columbian Hospital with all the investigating surgeons having adopted this practice in an attempt to prevent significant fracture collapse and neck shortening. Anecdotally, the investigators have not seen significant rates of cephalic screw cut-out over the past five years, and believe the investigators' screw cut-out rates are lower than what is reported in the literature. The investigators have been using the Gamma Nail (Stryker) to statically lock the screw as the previous TFN lacked the ability for static locking. However, with the advent of the TFN-A, the investigators have adopted this implant as their long cephalomedullary nail of choice for fixation of pertrochanteric femur fractures.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age
* AO/OTA 31-A fractures who the surgeon deems eligible for treatment with a cephalomedullary nail
* Open and closed fractures
* Ambulatory prior to injury (with or without walking aides)
* Native (non-fractured, no implant) contralateral hip
* Willing and able to sign consent (substitute decision maker)

Exclusion Criteria:

* Contralateral hip fracture or hip arthroplasty
* Fracture not amenable to treatment with a cephalomedullary nail
* Non-ambulatory patient
* Fractures >14 days (time of injury to OR)
* Bilateral pertrochanteric hip fractures
* Non-unions
* Pathologic fractures
* Periprosthetic fractures
* Patients with spinal injury
* Incarceration
* Pregnancy
* Limited life expectancy due to significant medical co-morbidities or medical contra-indications to surgery
* Likely problems, in the judgement of the investigators, with maintaining follow-up (i.e., patients with no fixed address, report a plan to move out of town, or intellectually challenged patients without adequate family support).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2021-05-17 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Radiographic Assessment | 12 months post treatment
  The primary objective of this study will be to investigate how statically locking the TFN-A influences shortening or collapse of pertrochanteric fractures by measuring radiographic shortening or collapse of pertrochanteric fractures treated with the TFN-A implant.

SECONDARY OUTCOMES:
Fracture Reduction Quality | Intra-operatively
  Assessed through x-rays of the entire proximal femur
Femoral Offset | 1 day post-op, 6 weeks, 12 weeks, 6 months, and 12 months
  Measured in a method described by O. Paul et al
Tip-Apex distance | 1 day post-op, 6 weeks, 12 weeks, 6 months, and 12 months
  Measured as described by Baumgaertner et al
Complications | intra-operatively, 1 day post-op, 6 weeks, 12 weeks, 6 months, and 12 months
  SAEs/AEs

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Perey, MD, FRCSC, Principal Investigator — Royal Columbian Hospital/Fraser Health Authority; David Cinats, MD, Principal Investigator — Orthopaedic Surgeon, Fraser Health Authority
Locations (1):
- Royal Columbian Hospital/Fraser Health Authority, New Westminster, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
Participant data will be kept confidential. Study findings and de-identified study data will be available to other researchers in the form of a published paper.

REFERENCES:
- [Background] Kanis JA, Oden A, McCloskey EV, Johansson H, Wahl DA, Cooper C; IOF Working Group on Epidemiology and Quality of Life. A systematic review of hip fracture incidence and probability of fracture worldwide. Osteoporos Int. 2012 Sep;23(9):2239-56. doi: 10.1007/s00198-012-1964-3. Epub 2012 Mar 15. PMID 22419370
- [Background] Zickel RE. A new fixation device for subtrochanteric fractures of the femur: a preliminary report. Clin Orthop Relat Res. 1967 Sep-Oct;54:115-23. No abstract available. PMID 5589594
- [Background] Stapert JW, Geesing CL, Jacobs PB, de Wit RJ, Vierhout PA. First experience and complications with the long Gamma nail. J Trauma. 1993 Mar;34(3):394-400. doi: 10.1097/00005373-199303000-00015. PMID 8483181
- [Background] Lecerf G, Fessy MH, Philippot R, Massin P, Giraud F, Flecher X, Girard J, Mertl P, Marchetti E, Stindel E. Femoral offset: anatomical concept, definition, assessment, implications for preoperative templating and hip arthroplasty. Orthop Traumatol Surg Res. 2009 May;95(3):210-9. doi: 10.1016/j.otsr.2009.03.010. Epub 2009 May 6. PMID 19423418
- [Background] Paul O, Barker JU, Lane JM, Helfet DL, Lorich DG. Functional and radiographic outcomes of intertrochanteric hip fractures treated with calcar reduction, compression, and trochanteric entry nailing. J Orthop Trauma. 2012 Mar;26(3):148-54. doi: 10.1097/BOT.0b013e31821e3f8c. PMID 21918483
- [Background] Yoo JH, Kim TY, Chang JD, Kwak YH, Kwon YS. Factors influencing functional outcomes in united intertrochanteric hip fractures: a negative effect of lag screw sliding. Orthopedics. 2014 Dec;37(12):e1101-7. doi: 10.3928/01477447-20141124-58. PMID 25437085
- [Background] Gausden EB, Sin D, Levack AE, Wessel LE, Moloney G, Lane JM, Lorich DG. Gait Analysis After Intertrochanteric Hip Fracture: Does Shortening Result in Gait Impairment? J Orthop Trauma. 2018 Nov;32(11):554-558. doi: 10.1097/BOT.0000000000001283. PMID 30239477
- [Background] Bishop JA, Palanca AA, Bellino MJ, Lowenberg DW. Assessment of compromised fracture healing. J Am Acad Orthop Surg. 2012 May;20(5):273-82. doi: 10.5435/JAAOS-20-05-273. PMID 22553099